CLINICAL TRIAL: NCT03299686
Title: A Randomized, Subject- and Investigator-blinded, Placebo Controlled, Multi-center, Multiple Dose Study to Assess the Efficacy and Safety of CJM112 in Patients With Inadequately Controlled Moderate to Severe Asthma
Brief Title: Study to Assess the Efficacy and Safety of CJM112 in Patients With Inadequately Controlled Severe Asthma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CCJM112X2204
Record Dates: First submitted 2017-08-07; First posted 2017-10-03 (Actual); Results first posted 2020-08-06 (Actual); Last update posted 2021-10-08 (Actual); Status verified 2021-10

CONDITIONS: Asthma
Keywords: Asthma, allergic, eosinophilic, non-T2 high, allergy triggered asthma, reactive asthma, asthma attack, difficulty breathing
MeSH Terms: conditions — Asthma; Dyspnea

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- CJM112 (Experimental): Study treatment
  Interventions: Drug: CJM112
- Placebo to CJM112 (Placebo Comparator): Placebo
  Interventions: Other: Placebo to CJM112

INTERVENTIONS:
Drug: CJM112 — 300 mg CJM112 (Study treatment) s.c. injection received per week for the first 4 weeks, followed by once every two weeks up to Week 12 (Day 85) + standard of care treatment.
  Arms: CJM112
Other: Placebo to CJM112 — Placebo to match CJM112 + standard of care treatment
  Arms: Placebo to CJM112

SUMMARY:
An unmet medical need exists for patients with moderate and severe asthma who continue to demonstrate symptoms despite being on standard of care medications, and are not eligible for other biologic therapies developed or in development for T2-high(allergic/eosinophilic) asthma. The purpose of this study was to determine if CJM112, an anti-IL-17A antibody, displayed the clinical efficacy and safety profile to support further development in patients with inadequately controlled moderate to severe asthma with low IgE and low circulating eosinophil levels.

DETAILED DESCRIPTION:
After an initial screening visit, run-in period and baseline assessments, the eligible subjects entered the treatment period and were randomized in a 3:2 ratio to one of the two treatment groups:

* 300 mg CJM112 s.c. injection received once per week for the first 4 weeks, followed by once every two weeks up to Week 12 (Day 85) + standard of care treatment.
* Matching placebo + standard of care treatment. After completion of the last dose on Day 85 of treatment period, subjects returned for the final efficacy assessment on Day 92. Following the treatment period, all subjects entered a 13-week safety follow-up period, including the End of Study (EoS) visit on Day 176.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with a physician-diagnosed history of moderate to severe asthma for a period of at least one year prior to screening.
2. Patients on a stable therapy regimen of asthma for at least 3 months prior to screening with at least medium dose inhaled glucocorticoid and at least one additional asthma controller medication (such as inhaled long-acting bronchodilator, leukotriene antagonist, theophylline, stable low dose glucocorticoid, etc).
3. Acceptable and reproducible spirometry with FEV1 ≥ 40 and ≤ 90% of predicted at screening and baseline (re-testing is allowed once).
4. ACQ score ≥ 1.5 at screening and baseline (re-testing is allowed once).
5. Total serum IgE < 150 IU/mL
6. Peripheral blood eosinophils <300/μL

Exclusion Criteria:

1. Previous use of biologics or other concomitant medications within the time periods specified in the SOM/protocol.
2. History of ongoing, chronic, or recurrent moderate or severe infectious disease.
3. Patients who have smoked or inhaled nicotine or tobacco products within the 6 month period prior to Visit 1 or who have a smoking history of greater than 10 pack years.
4. Patients who have had an asthma attack/exacerbation requiring systemic corticosteroids for at least 3 continuous days within 4 weeks prior to screening.
5. Patients who have had a respiratory tract infection or asthma worsening within 4 weeks prior to Visit 1 or during the screening period.
6. Women of child-bearing potential unless they use highly effective methods of contraception during dosing and for 13 weeks after stopping of investigational drug.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 118 (Actual)
Dates: Start 2017-11-06 (Actual); Primary Completion 2019-04-08 (Actual); Study Completion 2019-07-08 (Actual)

CONTACTS AND LOCATIONS:
Locations (27):
- United States (8):
  - Novartis Investigative Site, Fullerton, California
  - Novartis Investigative Site, Riverside, California
  - Novartis Investigative Site, Denver, Colorado
  - Novartis Investigative Site, Boston, Massachusetts
  - Novartis Investigative Site, St Louis, Missouri
  - Novartis Investigative Site, Raleigh, North Carolina
  - Novartis Investigative Site, Medford, Oregon
  - Novartis Investigative Site, Spartanburg, South Carolina
- Argentina (2):
  - Novartis Investigative Site, Mar del Plata, Buenos Aires
  - Novartis Investigative Site, Santa Fe, Rosario
- Belgium (3):
  - Novartis Investigative Site, Jette, Brussels Capital
  - Novartis Investigative Site, Ghent
  - Novartis Investigative Site, Liège
- Denmark (4):
  - Novartis Investigative Site, Aalborg
  - Novartis Investigative Site, Copenhagen NV
  - Novartis Investigative Site, Hvidovre
  - Novartis Investigative Site, Odense C
- France (2):
  - Novartis Investigative Site, Montpellier, Herault
  - Novartis Investigative Site, Lyon
- Germany (4):
  - Novartis Investigative Site, Berlin
  - Novartis Investigative Site, Großhansdorf
  - Novartis Investigative Site, Mainz
  - Novartis Investigative Site, Wiesbaden
- Israel (2):
  - Novartis Investigative Site, Jerusalem
  - Novartis Investigative Site, Rehovot
- Slovakia (2):
  - Novartis Investigative Site, Levice
  - Novartis Investigative Site, Spišská Nová Ves

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com

REFERENCES:
- See also: A Plain Language Trial Summary is available on novartisclinicaltrials.com — https://www.novctrd.com/ctrdweb/patientsummary/patientsummaries?patientSummaryId=599

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were from Argentina (2), Belgium (3), Germany (5), Denmark (4), France (2), Israel (3), Slovakia (2), The United States (7)
Pre-assignment Details: After an initial screening visit, run-in period and baseline assessments, the eligible subjects entered the treatment period and were randomized in a 3:2 ratio to one of the two treatment groups.
Groups:
- CJM112 300 mg: Study treatment: 300 mg CJM112 s.c. injection received once per week for the first 4 weeks, followed by once every two weeks up to Week 12
- Placebo: Placebo to CJM112: Placebo s.c. injection received once per week for the first 4 weeks, followed by once every two weeks up to Week 12
Period: Treatment Epoch
Arm/Group | CJM112 300 mg | Placebo
Started | 70 | 48
PD (Pharmacodynamics) Analysis Set (All subjects with available PD data, who received any study drug, and no major protocol deviations) | 69 | 48
Completed | 59 | 44
Not Completed | 11 | 4
Not completed — Subject/Guardian Decision | 2 | 0
Not completed — Physician Decision | 1 | 0
Not completed — Adverse Event | 8 | 4
Period: Follow-up Epoch
Arm/Group | CJM112 300 mg | Placebo
Started | 59 | 44
Completed | 59 | 43
Not Completed | 0 | 1
Not completed — Subject/Guardian Decision | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | CJM112 300 mg | Placebo | Total
Number analyzed (Participants) | 70 | 48 | 118
Age, Continuous [Mean (Standard Deviation); unit: Years] | 57.1 (12.79) | 55.9 (11.62) | 56.6 (12.29)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 39 | 32 | 71
  Male | 31 | 16 | 47
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 2 | 0 | 2
  Black or African American | 6 | 1 | 7
  Other | 1 | 0 | 1
  White | 61 | 47 | 108

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Forced Expiratory Volume in One Second (FEV1)
Description: The primary efficacy analysis assessed the effect of CJM112 on the absolute change from baseline in trough FEV1 in Liters compared to placebo on Day 92. Forced Expiratory Volume in one second (FEV1) is calculated as the volume of air forcibly exhaled in one second as measured by a spirometer. Baseline measurement was defined as the baseline visit pre-bronchodilator spirometry assessment.
Time Frame: Baseline, Day 92
Population: The analysis population included the Pharmacodynamics (PD) analysis set with evaluable FEV1 data at both timepoints.
Measure: Mean (Standard Deviation); unit: Liters
Arm/Group | CJM112 300 mg | Placebo
Number analyzed (Participants) | 53 | 36
Liters | 0.043 (0.031) | 0.016 (0.030)
Statistical Analysis 1: Comparison: CJM112 300 mg vs Placebo; Test type: Superiority; p = 0.7374, Bayesian linear repeated measures model — Probability CJM112 better than placebo; Mean Difference (Net) = 0.027, 80% CI 2-sided [-0.029 to 0.082], Standard Deviation 0.043; Lower limit and upper limit represents the Credibility Interval from the Bayesian analysis

2. Secondary Outcome: Change From Baseline in Forced Expiratory Volume 1 (FEV1) % of Predicted
Description: The secondary efficacy analyses assessed the effect of CJM112 on the absolute change from baseline in trough FEV1 in % of predicted compared to placebo on Day 92. Forced Expiratory Volume in one second (FEV1) was calculated as the volume of air forcibly exhaled in one second as measured by a spirometer. FEV1% of predicted is defined as FEV1% of the patient divided by the average FEV1% in the population for any person of similar age, sex and body composition. Pre-bronchodilator FEV1% of predicted was directly provided as part of the spirometry assessment.
Time Frame: Baseline, Day 92
Population: The analysis population included the Pharmacodynamics (PD) analysis set with evaluable FEV1 data at both timepoints
Measure: Least Squares Mean (Standard Error); unit: Percent predicted
Arm/Group | CJM112 300 mg | Placebo
Number analyzed (Participants) | 53 | 36
Percent predicted | 1.064 (0.914) | 0.151 (1.105)
Statistical Analysis 1: Comparison: CJM112 300 mg vs Placebo; Test type: Superiority; p = 0.263, Mixed Models Analysis — 1-sided p-value; p-value smaller than 0.1 is considered as statistically significant; Mean Difference (Net) = 0.913, 80% CI 2-sided [-0.939 to 2.766], Standard Error of Mean 1.434

3. Secondary Outcome: Change From Baseline in Asthma Control Questionnaire 6 (ACQ6) Score
Description: The ACQ-6 is a validated asthma assessment tool that consists of 6 self-assessment questions. Each item on the ACQ-6 has a possible score ranging from 0 to 6 and the total score is the mean of all responses. The seven-point response scale goes from 0 = 'totally controlled' to 6 = 'severely uncontrolled.
  Negative change from baseline values indicate improved asthma control.
Time Frame: Baseline, Day 92
Population: The analysis population included the Pharmacodynamics (PD) analysis set with evaluable ACQ6 data at both timepoints
Measure: Least Squares Mean (Standard Error); unit: units on scale
Arm/Group | CJM112 300 mg | Placebo
Number analyzed (Participants) | 56 | 41
units on scale | -0.93 (0.09) | -0.71 (0.11)
Statistical Analysis 1: Comparison: CJM112 300 mg vs Placebo; Test type: Superiority; p = 0.061, Mixed Models Analysis — 1-sided p-value; p-value smaller than 0.1 is considered as statistically significant; Mean Difference (Net) = -0.22, 80% CI 2-sided [-0.41 to -0.04], Standard Error of Mean 0.14

4. Secondary Outcome: Change From Baseline in Asthma Control Questionnaire 7 (ACQ7) Score
Description: The ACQ-7 measured asthma symptom control and consists of 7 items: 5 on symptom assessment, 1 on rescue medication use and 1 on airway calibre (FEV1 % predicted). All seven items are scored on a 7-point Likert scale, with 0 indicating total control and 6 indicating poor control. The questions are equally weighted and the total score is the mean of the seven items. The first 6 questions of the ACQ-7 were completed by the participant while the last question was completed by the study investigator using data from the Master Scope spirometer. A negative change from baseline indicates improvement in lung function.
Time Frame: Baseline, Day 92
Population: The analysis population included the Pharmacodynamics (PD) analysis set with evaluable ACQ7 data at both timepoints
Measure: Least Squares Mean (Standard Error); unit: units on scale
Arm/Group | CJM112 300 mg | Placebo
Number analyzed (Participants) | 53 | 36
units on scale | -0.83 (0.08) | -0.60 (0.10)
Statistical Analysis 1: Comparison: CJM112 300 mg vs Placebo; Test type: Superiority; p = 0.040, Mixed Models Analysis — 1-sided p-value; p-value smaller than 0.1 is considered as statistically significant; Mean Difference (Net) = -0.23, 80% CI 2-sided [-0.40 to -0.06], Standard Error of Mean 0.13

5. Secondary Outcome: Percentage of Patients With at Least 0.5 Decrease in ACQ7 Score
Description: The ACQ-7 measured asthma symptom control and consists of 7 items: 5 on symptom assessment, 1 on rescue medication use and 1 on airway calibre (FEV1 % predicted). All seven items are scored on a 7-point Likert scale, with 0 indicating total control and 6 indicating poor control. The questions are equally weighted and the total score is the mean of the seven items. The first 6 questions of the ACQ-7 were completed by the participant while the last question was completed by the study investigator using data from the Master Scope spirometer. A negative change from baseline indicates improvement in lung function.
  An ACQ7 responder is defined as a patient with a decrease in score of greater or equal to 0.5 when compared to baseline.
Time Frame: Baseline, Day 92
Population: The analysis population included the Pharmacodynamics (PD) analysis set with evaluable ACQ7 data at both timepoints
Measure: Count of Participants; unit: Participants
Arm/Group | CJM112 300 mg | Placebo
Number analyzed (Participants) | 53 | 36
Participants | 38 | 19

6. Secondary Outcome: Percentage of Patients With Adverse Events (AEs) Leading to Discontinuation of Study Treatment
Description: Number of patients with at least one adverse event leading to discontinuation of study treatment
Time Frame: 85 days
Population: Safety analysis set: Subjects who received any study drug
Measure: Count of Participants; unit: Participants
Arm/Group | CJM112 300 mg | Placebo
Number analyzed (Participants) | 70 | 48
Participants | 8 | 4

ADVERSE EVENTS:
Time Frame: Adverse events were collected from first dose of study treatment until end of study treatment plus 91 days post treatment, up to maximum duration of 6 months
Description: Any sign or symptom that occurs during the study treatment plus the 91 days post treatment
Arm/Group | CJM112 300 mg | Placebo
All-Cause Mortality (participants affected / at risk) | 0/70 | 0/48
Serious Adverse Events (participants affected / at risk) | 3/70 | 2/48
Other Adverse Events (participants affected / at risk) | 55/70 | 38/48
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | CJM112 300 mg (N=70) | Placebo (N=48)
Stress cardiomyopathy (Cardiac disorders) | 0 | 1
Asthenia (General disorders) | 1 | 0
Pneumonia (Infections and infestations) | 0 | 1
Urinary tract infection (Infections and infestations) | 1 | 0
Depression (Psychiatric disorders) | 1 | 0
Asthmatic crisis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | CJM112 300 mg (N=70) | Placebo (N=48)
Arrhythmia supraventricular (Cardiac disorders) | 0 | 1
Hypothyroidism (Endocrine disorders) | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 1
Constipation (Gastrointestinal disorders) | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 3 | 3
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 2 | 1
Nausea (Gastrointestinal disorders) | 3 | 2
Proctalgia (Gastrointestinal disorders) | 0 | 1
Toothache (Gastrointestinal disorders) | 1 | 1
Vomiting (Gastrointestinal disorders) | 0 | 2
Asthenia (General disorders) | 0 | 1
Fatigue (General disorders) | 4 | 3
Injection site haematoma (General disorders) | 1 | 1
Oedema peripheral (General disorders) | 1 | 1
Pyrexia (General disorders) | 1 | 1
Bronchitis (Infections and infestations) | 5 | 3
Conjunctivitis (Infections and infestations) | 0 | 1
Cystitis (Infections and infestations) | 2 | 1
Gastroenteritis (Infections and infestations) | 2 | 1
Gastroenteritis viral (Infections and infestations) | 0 | 1
Lower respiratory tract infection (Infections and infestations) | 2 | 0
Nasopharyngitis (Infections and infestations) | 16 | 6
Oral candidiasis (Infections and infestations) | 4 | 0
Oral herpes (Infections and infestations) | 0 | 1
Pharyngitis (Infections and infestations) | 1 | 2
Respiratory tract infection (Infections and infestations) | 2 | 1
Respiratory tract infection viral (Infections and infestations) | 2 | 1
Rhinitis (Infections and infestations) | 0 | 1
Sinusitis (Infections and infestations) | 3 | 0
Tooth abscess (Infections and infestations) | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 4 | 2
Urinary tract infection (Infections and infestations) | 1 | 2
Viral upper respiratory tract infection (Infections and infestations) | 2 | 1
Arthropod sting (Injury, poisoning and procedural complications) | 0 | 1
Fall (Injury, poisoning and procedural complications) | 0 | 1
Ligament sprain (Injury, poisoning and procedural complications) | 0 | 1
Rib fracture (Injury, poisoning and procedural complications) | 0 | 1
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 | 1
Subcutaneous haematoma (Injury, poisoning and procedural complications) | 0 | 1
Alanine aminotransferase increased (Investigations) | 0 | 2
Amylase increased (Investigations) | 0 | 1
Aspartate aminotransferase increased (Investigations) | 0 | 1
Blood alkaline phosphatase increased (Investigations) | 0 | 1
Blood bicarbonate decreased (Investigations) | 0 | 1
Blood cholesterol increased (Investigations) | 1 | 1
Blood creatine phosphokinase increased (Investigations) | 1 | 1
Blood creatinine increased (Investigations) | 1 | 1
Blood lactate dehydrogenase increased (Investigations) | 1 | 1
Blood potassium increased (Investigations) | 0 | 1
Blood triglycerides increased (Investigations) | 0 | 1
Gamma-glutamyltransferase increased (Investigations) | 0 | 1
Lipase increased (Investigations) | 0 | 1
Protein urine present (Investigations) | 0 | 1
Red blood cell sedimentation rate increased (Investigations) | 0 | 1
Gout (Metabolism and nutrition disorders) | 0 | 1
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 3 | 5
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 | 1
Limb discomfort (Musculoskeletal and connective tissue disorders) | 2 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 | 0
Dizziness (Nervous system disorders) | 4 | 0
Headache (Nervous system disorders) | 8 | 6
Intercostal neuralgia (Nervous system disorders) | 0 | 1
Migraine (Nervous system disorders) | 2 | 0
Sciatica (Nervous system disorders) | 0 | 1
Insomnia (Psychiatric disorders) | 0 | 1
Prostatitis (Reproductive system and breast disorders) | 0 | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 16 | 13
Cough (Respiratory, thoracic and mediastinal disorders) | 4 | 4
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 3 | 3
Rash (Skin and subcutaneous tissue disorders) | 1 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (ie, data from all sites) in the clinical trial.

DOCUMENTS (2):
  • Study Protocol (2018-05-15): https://cdn.clinicaltrials.gov/large-docs/86/NCT03299686/Prot_001.pdf
  • Statistical Analysis Plan (2019-08-14): https://cdn.clinicaltrials.gov/large-docs/86/NCT03299686/SAP_000.pdf